CLINICAL TRIAL: NCT04988126
Title: Assessment of Pain, Fatigue and Quality of Life in COVID-19 Patients
Brief Title: Pain, Fatigue and Life Quality in COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Ali İzzet Akçin, Research Assistant-MD, Afyonkarahisar Health Sciences University
Other Study IDs: SAA21Covid19
Record Dates: First submitted 2021-07-29; First posted 2021-08-03 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Pneumonia; Pain; Fatigue; Quality of Life
Keywords: COVID-19 Pneumonia; Pain; Fatigue; Quality of Life
MeSH Terms: conditions — Pain; Fatigue | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Group: Patient with Covid 19 Pneumonia
  Interventions: Other: Interventions

INTERVENTIONS:
Other: Interventions — Observational study, not applicable

SUMMARY:
The aim in this study is to evaluate pain, fatigue and quality of life in patients with Covid-19 pneumonia in long-term follow-up and to investigate their relationship with pneumonia severity, age, presence of comorbidity and depression level.

DETAILED DESCRIPTION:
Patients over the age of 18 who are hospitalized in the Pandemic Service, and are positive for COVID-19 PCR, will be included in the study if the participants read the informed consent form and volunteer for the study.

Patients' age, comorbidities, initial symptoms, and pneumonia severity (mild/moderate/severe) will be recorded. Pain, fatigue and depression assessments will be made on the first day of hospitalization, at discharge, at the 1st month and 3rd month after discharge. The 1st and 3rd month evaluations of the patients will be made by contacting the participants by phone. In addition to the 1st and 3rd month evaluations, the quality of life will also be evaluated with the SF-12 questionnaire.

ELIGIBILITY:
Inclusion Criteria: Patients over the age of 18 who are hospitalized in the Pandemic Service, and are positive for COVID-19 PCR, will be included in our study.

* Patient with Covid 19 Pneumonia

Exclusion Criteria:

* Uncooperative Patient,
* Illiterate Patients,
* Pregnancy,
* Patients with Chronic Pain or Fatigue in the last 6 months (before COVID-19 disease),
* Patients who were admitted to the intensive care unit during their hospitalization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who are hospitalized in the Pandemic Service, and are positive for COVID-19 PCR
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | up to 12th week
  Change from baseline visual analog scale (VAS) myalgia, arthralgia, cervical, thorocic and lumbar pain at 4th and 12th week.
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

SECONDARY OUTCOMES:
Fatigue Severity Scale | up to 12th week
  The scale evaluates the fatigue severity of the participants in the last week. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. The minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities.
Hospital Anxiety And Depression Scale | up to 12th week
  The Hospital Anxiety and Depression Scale (HADS) is a measure designed to assess anxiety and depression symptoms in patients. The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. A subscore of > 7 for depression and > 10 for anxiety would indicate a clinical case.
Short form 12 (SF-12) | up to 12th week
  The SF-12 is an easy-to-administer questionnaire with proven reliability and validity, obtained by shortening and simplifying the SF-36. It is used in the assessment of physical and mental health, the two main components of general health. SF-12 surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning

CONTACTS AND LOCATIONS:
Overall Officials: Sevda MD ADAR, Principal Investigator — Afyonkarahisar Health Sciences University; Ali İzzet MD AKÇİN, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cipollaro L, Giordano L, Padulo J, Oliva F, Maffulli N. Musculoskeletal symptoms in SARS-CoV-2 (COVID-19) patients. J Orthop Surg Res. 2020 May 18;15(1):178. doi: 10.1186/s13018-020-01702-w. No abstract available. PMID 32423471
- [Background] Garrigues E, Janvier P, Kherabi Y, Le Bot A, Hamon A, Gouze H, Doucet L, Berkani S, Oliosi E, Mallart E, Corre F, Zarrouk V, Moyer JD, Galy A, Honsel V, Fantin B, Nguyen Y. Post-discharge persistent symptoms and health-related quality of life after hospitalization for COVID-19. J Infect. 2020 Dec;81(6):e4-e6. doi: 10.1016/j.jinf.2020.08.029. Epub 2020 Aug 25. PMID 32853602
- [Background] Halpin SJ, McIvor C, Whyatt G, Adams A, Harvey O, McLean L, Walshaw C, Kemp S, Corrado J, Singh R, Collins T, O'Connor RJ, Sivan M. Postdischarge symptoms and rehabilitation needs in survivors of COVID-19 infection: A cross-sectional evaluation. J Med Virol. 2021 Feb;93(2):1013-1022. doi: 10.1002/jmv.26368. Epub 2020 Aug 17. PMID 32729939